CLINICAL TRIAL: NCT00966784
Title: The Effect of 2 Months Daily Supplementation of Orange Juice With Fibers
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Responsible Party: Tel-Aviv Sourasky Medical Center
Other Study IDs: TASMC-09-NV-233-CTIL
Record Dates: First submitted 2009-08-26; First posted 2009-08-27 (Estimated); Last update posted 2009-08-27 (Estimated); Status verified 2009-08

CONDITIONS: Healthy People
MeSH Terms: interventions — Dietary Fiber

INTERVENTIONS:
Other: Dietary Fibers

SUMMARY:
The study hypothesis is that 2 Months Daily Supplementation of Orange juice with fibers will effect the weight and the plasma lipids.

This will be a double-blind parallel controlled study. Study population will include 50 subjects, who will be divided randomly into two groups. The first group will get the Orange juice with fibers, and the second group will get Orange juice with out the fibers.

ELIGIBILITY:
Inclusion Criteria:

* Healthy Volunteers
* Age 60>18 years
* Written informed consent
* Consumers of orange drinks: freshly squeezed juices, commercial pasteurized juices and / or orange soft drinks
* Regular eating pattern

Exclusion Criteria:

* Patients with chronic disease sach as:

  * diabetes,
  * cancer,
  * C.O.P.D.,
  * metabolic syndrome,
  * over weight,
  * kidney failure,
  * heart disease and
  * osteoporosis.
* Antibiotic treatment in the last 4 weeks
* Subjects on regular probiotic or prebiotic supplementation, unless the subject will do 2 weeks of wash out before commencing the study.
* Subjects with intestinal disorders such as: IBD, IBS, celiac, colon cancer.
* Subjects after intestinal surgery.
* Use of medicines for lowering cholesterol (simvastatin), sugar control
* Pregnancy
* Subjects with abnormal base-line blood test results: liver functions and/or kidney functions, cholesterol level above 200 mg/dL and glucose level above 50 mg/dL (during fast)

Ages: 18 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2009-09; Primary Completion 2010-09 (Estimated); Study Completion 2010-12 (Estimated)

PRIMARY OUTCOMES:
To examine the effect of 2 Months Daily Supplementation of Orange Juice with fibers on the weight and the plasma lipids

CONTACTS AND LOCATIONS:
Locations (1):
- Suorasky Medical Center, Tel Aviv, Israel